CLINICAL TRIAL: NCT07132372
Title: The Role of Birth Memories in the Relationship Between Maternal Functioning and Blues
Acronym: Birth
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ece Kaplan, Asisstant Professor Obstetrics and Gynecology Nursing, University of Gaziantep
Other Study IDs: GAUN-EBE-EKD-03
Record Dates: First submitted 2025-07-25; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-06

CONDITIONS: Women (Between 18 to 50 Years Old)
Keywords: Maternal function; maternity blues; birth memory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data were collected using a personal information form, BIMF, PMBAS, and BirthMARQ.: Data were collected using a personal information form, BIMF, PMBAS, and BirthMARQ.
  Interventions: Other: Birth Memories and Recall scale

INTERVENTIONS:
Other: Birth Memories and Recall scale — The data collection tools were applied to the participants by the researcher through face-to-face interviews. At the outset, the purpose of the study was explained to the participants. It was stated that participation in the study was completely voluntary and that they could withdraw from the study at any time. Then, their written and verbal consent was obtained.Participants who agreed to participate in the study, had no condition that would prevent communication, and had babies between the ages of 0 and 1 were included in the study.Data were collected using a personal information form, BIMF, PMBAS, and BirthMARQ.

SUMMARY:
This study was conducted to examine role of birth memories and recall in relationship between maternal functioning and maternity blues in postpartum women.A cross-sectional design was employed. The study sample consisted of 418 participants from this population.

DETAILED DESCRIPTION:
The sustainability of postpartum maternal functioning has increasingly attracted attention in the literature in terms of how the birth experience is cognitively processed and the possible effects of the way it is recalled on maternity blues. This study was conducted to examine the role of birth memories and recall in relationship between maternal functioning and maternity blues in postpartum women.A cross-sectional design was employed. The study sample consisted of 418 participants from this population. Data were collected using a personal information form, Barkin Index of Maternal Functioning , Postpartum Maternity Blues Assessment Scale and Birth Memories and Recall Questionnaire .

ELIGIBILITY:
Inclusion Criteria:

* Mothers with babies aged 0-1 who volunteered to participate in the study who had no conditions that would prevent communication.

Exclusion Criteria:

* Mothers with babies over 1 year old who do not wish to participate in the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study consisted of mothers who presented to the pediatrics outpatient clinic of the hospital between May 30 and August 30, 2024 and had babies between the ages of 0 and 1. The G*Power software was used to calculate the sample size. Previous studies were examined (Oruç & Kukulu, 2022; Kılıç Doğan & Cesur, 2023) and the expected confidence intervals of the Barkin Index of Maternal Functioning were determined. Accordingly, the sample size was calculated as 90 participants, based on a confidence interval of α = 0.05, a test power (1-β) of 0.95, and an effect size of dz = 0.306. Eventually, the study was completed with 418 participants.
Sampling Method: Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
The Barkin Index of Maternal Functioning | 3 months
  The study was completed with 418 participants. Their written and verbal consent was obtained.
  The Barkin Index of Maternal Functioning: The scale consists of 16 seven-point Likert items.The lowest score from the scale is 0, and the highest is 96. The higher the score is, the higher the functioning is.
The Postpartum Maternity Blues Assessment Scale | 3 months
  The Postpartum Maternity Blues Assessment Scale: It has 23 five-point Likert items. The total scores range from 23 to 115. A high score indicates that symptoms of maternity blues are high in the postpartum period.
The Birth Memories and Recall Questionnaire | 3 months
  The Birth Memories and Recall Questionnaire: The scale consists of a total of 21 items and 6 sub-dimensions. The mean score of the items on each sub-dimension gives the sub-dimension score. Items 1, 3, and 11 are reverse-scored. The total scores range from 27 to 189. The higher the score is, the higher the memories is. The sub-dimensions are emotional memory, ambivalent emotional memory, centrality of memory, coherence and reliving, sensory memory, and involuntary recall.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Kaplan doğan, Dr., Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Maternal and paternal postpartum early mood and bonding — https://pubmed.ncbi.nlm.nih.gov/36593232/